CLINICAL TRIAL: NCT06429189
Title: An Online Home-based Combined Exercise Intervention With Self-selected Intensity for Women With Breast Cancer: The Home-Combo Randomized Controlled Trial.
Brief Title: Home-Combo: an Online Home-based Combined Exercise Intervention for Women With Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Lusófona (Other)
Collaborators: Universidade Lusófona de Humanidades e Tecnologias (Other); Grupo HPA (Unknown); Associação Oncológica do Algarve (Unknown); Liga Portuguesa Contra o Cancro (Unknown); Centro Hospitalar Universitario do Algarve (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Home-Combo
Record Dates: First submitted 2024-05-03; First posted 2024-05-24 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Chemotherapy Effect
Keywords: Breast cancer; Home-based exercise; Functional performance; Body composition; Physical activity; Quality of life
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: 2-arm pragmatic and superiority randomized controlled trial with an intervention and an active control group, with a 1:1 allocation ratio.
  Participants in this group will perform a home-based combined exercise program throughout their chemotherapy treatments, starting within 1-2 weeks of its start and ending within 3-4 weeks post-treatment completion.
  Women randomized to the control group will receive weekly 30-minute supervised sessions with breathing, stretching, relaxation exercises, and meditation during the intervention period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be told they are part of an exercise intervention without any mention of a control group.
  Healthcare professionals responsible for the chemotherapy prescription and administration and registering all clinical information will be blinded to the participants' groups.
  None of the research team members will know the number of participants, so data analysis will be performed in a blinded setting.
  If, at any given moment, a participant reveals her number to a research team member, all posterior data from that participant will be disregarded.
  If a participant decides to leave the study or must abandon it due to health complications, the team member with the number information will be informed, and data will be disregarded from the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based combined exercise (Experimental): Exercise intervention will be led by qualified exercise professionals online via Zoom. It will consist of two weekly 60-minute online exercise group sessions: a 5-minute warm-up, 30-minute resistance training, and a 20-minute aerobic exercise component, finishing with a 5-minute cooldown.
  The warm-up will consist of mobility and activation movements. The resistance training component will consist of 9 exercises involving large muscle groups, performed with body weight or free weights. The exercises will be completed in 2-3 sets of 10-15 repetitions. The aerobic component will consist of low-impact dance exercises that move large muscle groups to increase heart rate. The cooldown will consist of breathing exercises and light stretches.
  Interventions: Behavioral: Home-based combined exercise program with self-selected intensity
- Active control group (Placebo Comparator): The control group will receive weekly 30-minute supervised sessions with breathing, stretching, relaxation exercises, and meditation.
  Interventions: Behavioral: Home-based combined exercise program with self-selected intensity

INTERVENTIONS:
Behavioral: Home-based combined exercise program with self-selected intensity — Before the beginning of the exercise program, participants will receive an education session on how to use Borg's Perceived Rate of Exertion Scale (RPE) to monitor their effort during aerobic and resistance training and tips on when they may increase the exercise intensity. During the training sessions, participants in the intervention group will be asked to choose their preferred load to execute each exercise in the resistance component, told to perform the aerobic exercises at their preferred speed, and informed that they can stop exercising whenever they need to rest. The exercise professional may suggest increasing loads in specific exercises, but these increases will not be imposed on the participants. Attendance to the sessions in the intervention and control groups will be registered. Additionally, women in this group will be encouraged to perform brisk walking at their preferred intensity and receive a pedometer to increase walking motivation.
  Other Names: Home-combo

SUMMARY:
Background. Chemotherapy drugs carry many side effects that may hinder the functional performance of women with breast cancer (BC). Chemoresistance can lead to treatment failure. A relative dose intensity of chemotherapy <85% is associated with a worse diagnosis and lower treatment efficacy. Exercise may modulate treatment response through its effects on the tumor microenvironment and treatment tolerability. The need for a pleasant and sustainable exercise practice is important, considering the psychological and physiological stress that accompanies women with a BC diagnosis during treatment. Studies investigating the effects of exercise interventions on chemotherapy completion rates are needed.

Background. Chemotherapy drugs carry many side effects that may hinder the functional performance of women with breast cancer (BC). Chemoresistance can lead to treatment failure. A relative dose intensity of chemotherapy <85% is associated with a worse diagnosis and lower treatment efficacy. Exercise may modulate treatment response through its effects on the tumor microenvironment and treatment tolerability. The need for a pleasant and sustainable exercise practice is important, considering the psychological and physiological stress that accompanies women with a BC diagnosis during treatment. Studies investigating the effects of exercise interventions on chemotherapy completion rates are needed.

Purpose. This study will be a 2-arm pragmatic randomized controlled trial, Home-Combo, which will target Portuguese women with a breast cancer diagnosis undergoing either neo-adjuvant or adjuvant chemotherapy. The Home-Combo study primarily aims to investigate the effects of a structured, supervised, home-based combined exercise intervention with self-selected intensity, conducted across the chemotherapy treatment period, on the chemotherapy completion rates of women with BC. Secondly, this study intends to analyze the impact of this intervention on functional performance, body composition, PA levels, and quality of life. A 3-month follow-up will be performed to investigate short-term outcomes and active lifestyle sustainability post-intervention.

Methods. A 2-arm randomized controlled trial will be implemented in a real-world exercise setting to compare an online structured and supervised group aerobic and strength exercise intervention with an active control group during chemotherapy treatments. The study recruitment goal is 98 women with a BC diagnosis stage I-III who are scheduled to have neoadjuvant or adjuvant chemotherapy. Outcome measures will be obtained at baseline, mid-treatment (≈3 months), post-intervention (≈6 months), and 3-month follow-up. A mediation analysis will also be conducted.

Hypothesis 1: Women in the intervention will have a better completion rate than those in the control group.

Hypothesis 2: Women in the intervention will present better functional performance, body composition, PA levels, and quality of life than the control group.

Hypothesis 3: In the post-intervention period, women in the intervention group will maintain a more physically active lifestyle than women in the control group.

DETAILED DESCRIPTION:
Study setting The Home-Combo study will take place in the Algarve, and the sample will be recruited by medical referral from various public and private hospitals across the region.

The intervention design will consider the PA/exercise preferences, perceived barriers, and facilitators of women with BC. This information will be collected before the intervention through a mixed-methods qualitative study that will include a survey and focus groups. The intervention will be conducted online to ensure the participants' safety during the chemotherapy treatment phase, as they may have compromised immunity. Also, this option was made to attenuate participants' burden caused by commuting requirements. Participants will be enrolled in two cohorts.

Criteria for discontinuing or modifying allocated interventions Participants will be informed in the pre-study initial meeting that they may leave the study anytime. Participants will be asked to refrain from continuing the intervention if a worsening clinical condition prevents them from exercising and performing the assessments safely. The exercise program might be reviewed and tailored to the participants' condition across the intervention.

Strategies to improve adherence Before implementing this study, a survey and focus-group-based study will be performed to adjust the exercise program to the preferences, perceived barriers, and facilitators of women with a breast cancer diagnosis, considering the environmental and cultural context from where the intervention will be conducted. The supervising professional will monitor adherence to the supervised sessions through presence registration. This study will also consider the participants' adherence to the control group. To attempt dropout minimization, the investigators will have an active control group.

Concomitant care Physiotherapy treatments prescribed by the participant's primary physician and any exercises prescribed to be performed at home prescribed by the physiotherapist will be allowed during the intervention. Participants in the study will be asked not to engage in other exercise and PA programs or activities outside the program. Participants in the control group will not be prohibited from performing physical activities like brisk walking.

Sample size Considering this study design, sample size calculations were made for the primary outcome with a factorial variance analysis with repeated measures as reference statistical analysis, giving an initial estimation of 82 participants. Based on previous findings and considering a 20% dropout, the sample size was estimated at 98 participants with a moderate effect size (a=0.05; statistical power=0.80) according to Cohen's D calculations, using G* Power 3.1.

Recruitment Recruitment will occur through medical referrals from primary physicians of several public and private hospitals in the Algarve region. Additionally, the project will be presented at breast cancer-themed congresses and events, and digital flyers with information about the study will be made to assist in disseminating the project and the recruitment process. A research team member will then contact patients referred by the doctors to receive detailed information about the study. Optionally, patients can call the research team directly or contact them through email if they prefer. After confirming eligibility criteria and interest in participating in the study, patients will be asked to attend an initial session where more information will be given, and the informed consent will be signed. During that session, participants will be told they are not obliged to participate in the study and may decide to leave the project. Consent for data collection or sharing will also be obtained.

Data collection methods Assessments will be conducted in standardized conditions, in a clinical setting, in a calm and comfortable environment, in small groups, and performed by a qualified exercise professional. The assessments will be conducted in the morning, starting with the body composition measurements, followed by a 15-minute pause so participants can eat (since they will be weighted while fasting), preceded by a 10-minute warm-up with general movements to mobilize big muscle groups and the physical tests, that will be performed in the following order: shoulder angular measurements, strength, mobility, and aerobic endurance. Participants will be divided into small groups to facilitate instruction and conduction of the tests. Participants will receive the accelerometers one week before the field tests and return them on the physical assessment day. After the field measurements, all questionnaires will be delivered and answered through email (Google Forms)

Plans to promote retention The conducting exercise professional will control participants' adherence to the exercise program through a presence registry collected by the research team member with access to the list of participants' numbers. After the session, the non-interventionist research team member will pass the presence list to the respective numbers of the participants for program adherence analysis. If a participant fails to attend a session, contact will be made to ensure the participant's welfare and motivate them to participate in the next session. The data analysis will not consider participants who fail to attend 50% or more sessions. Positive feedback will be given to the participants during the sessions, as positive feedback enhances feelings of competence, enjoyment, and interest in the activity 86. Additionally, participants will be encouraged to keep an activity diary where they may register all activities performed autonomously. Participants will be contacted one week before the assessment to confirm their availability and presence. Data from participants who fail to perform the assessments during the intervention period will be excluded from data analysis. After the intervention, participants will be contacted monthly to check their well-being and keep their interest and motivation in engaging in the follow-up assessment.

Data management All the data collected in this study will be kept confidential, computerized, and encrypted in a database without any elements that may allow identification of the participants. After the participants have expressed interest and written informed consent, a number corresponding to the participant ID during the study will be provided. When the participant receives her ID number, all data inserted in the databases will not be directly linked to the participant's personal identification. A dataset will be created for each assessment time point. All datasets will be maintained by the members responsible for the investigation on a secure server of CIDEFES-UL for ten years and will be used exclusively for research purposes. Datasets used for specific analyses or to develop sub-studies will contain only the necessary variables and the demographical indicators provided to the research team members upon request to the leading investigator.

Statistical methods All data will be analyzed using IBM SPSS (version 29.0). Factorial ANCOVAS with repeated measures will be used for the primary and secondary outcomes, adjusted for potential covariates (e.g., concomitant treatments, BC diagnosis, neo-adjuvant/ adjuvant chemotherapy). Independent sample T-tests will be used to compare results between groups at each time point, considering chemotherapy completers versus non-completers. A Fisher's exact test will compare the proportion of participants who needed chemotherapy adjustments from those who did not. The intention-to-treat analysis will be conducted to ensure that all participants are included in the overall assessment, considering their compliance with the study protocol. The Last Observation Carried Forward method will be used to input missing data values. A per-protocol analysis will also be conducted without participants who failed to complete at least 50% of the training sessions. Normality plots and Kolmogorov-Smirnov tests will be performed to test the normality of outcome variables. If normality is not satisfied, non-parametric tests will be applied (e.g., Krustal-Wallis). Mediators of change (i.e., mechanisms by which RDI) will be explored using structural equation modeling (AMOS 18.0) and multiple mediation analysis (PROCESS macro for SPSS). Putative candidates will include treatment (e.g., dose planned vs. given dose, planned cycles minimum/maximum, treatment interruption ratios, response to treatment, percentage of participants who needed dose adjustments, and the mean value of dose adjustment), and physiological (e.g., body composition, functional performance, handgrip strength, PA levels) variables. Mediation occurs when a causal effect of an independent variable occurs on a dependent variable, partly or entirely explained by a mediator. Indirect effects testing will be performed using Preacher and Hayes' procedures.

Data monitoring A data monitoring committee will not be required for this trial as the interventions pose minimal risk, and participants will be protected by personal insurance throughout the study.

Harms All participants will have their adverse events monitored throughout the study, whether directly related to the intervention or not (if applicable). This monitoring will be done through self-reporting at the start of each session, registered for analysis and report purposes, or by their primary care physicians. Participants will be advised to contact the clinical team if they have difficulties.

Auditing Two authors will supervise all trial procedures and cross-check the interventionist actions and study processes. Additionally, an independent person external to the project will review the protocol.

Research ethics approval This study has received ethical approval from the collaborating hospital (UAIF 069/2024). This trial will follow the World Medical Association's Declaration of Helsinki for Human Studies.

Consent or assent Healthcare professionals will approach potential participants to determine if they are interested in participating. If they express interest, they will be referred to a research team member who will contact them. Additionally, interested participants will be allowed to share the study information with other women who have been diagnosed with breast cancer. If any of these women express interest in participating, they will also be considered after obtaining medical clearance. Once the eligibility criteria for the study are confirmed and the women express their interest in participating, they will receive the Informed Consent through email. In the informational session, women will be asked to digitally fill out and sign the Informed Consent. It will be clear to the participants that they can withdraw their consent anytime. After the informational session, a PDF copy of the signed Informed Consent will be emailed to each participant. The research team will also take additional measures to collect and share the participants' data.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer stage I-III diagnosis
* Scheduled to receive neoadjuvant or adjuvant chemotherapy
* Have acess to a computer

Exclusion Criteria:

* Medical conterindication to perform exercise or physical assessments due to concomitant comorbidity
* Non-controlled health conditions or diseases
* Psychological illness
* Currently enrolled in a structured exercise program
* Unable to complete the entire program (e.g., due to scheduled surgery or personal commitments)
* Pregnancy
* Worsening of clinical condition during intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 98 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy completion rates | Assessments will be performed at three time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months).
  The outcome will be reported as the mean RDI (mg.m-2/wk-1), which corresponds to a fraction of the planned chemotherapy dose intensity, by dividing the dose of chemotherapy per square meter (of surface area where the drug is related) in each cycle by the number of weeks in a cycle. Information regarding the planned chemotherapy treatment and the effectively received treatment (i.e., dose, type, and duration) will be acquired from medical records after signing the informed consent 53,19. Successful chemotherapy completion rate will be considered if the RDI is ≥85% of the planned treatment. Calculations to compare the actual chemotherapy dose intensity received and the initially planned dose intensity will be calculated as total milligrams of chemotherapy divided by the product of the body surface (in square meters) and total weeks of treatment. The RDI results from the actual dose intensity received are divided by the planned dose intensity.

SECONDARY OUTCOMES:
Functional performance | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  The 6-minute walk test will assess aerobic endurance, a standardized field test performed indoors in a 30-meter corridor with two turning points. Participants will be asked to walk the maximum distance possible.
Functional performance | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  Arm curls will assess upperbody strength. Participants will be instructed to perform as many repetitions as possible for 30 seconds with a 5-pound dumbbell.
Functional performance | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  Sit-to-stand tests assess lower body strength. Participants will be instructed to stand upright and sit entirely back on a chair as many times as possible within 30 seconds, maintaining their feet steady on the ground and the arms crossed with hands on the shoulders
Functional performance | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  Handgrip strength will be measured using a dynamometer and considered to the nearest 0.1kg. While performing the handgrip test for each hand, participants will be instructed to stand upright with feet at hip width and elbows completely stretched while applying the maximum grip continuously for more than 3 seconds.
Functional performance | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  Timed up-and-go tests will assess participants' overall mobility. Participants will be instructed to rise from a chair, walk 2.44 meters, turn around, walk back to the chair, and sit down.
Functional performance | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  A goniometer will perform shoulder flexion and abduction angular measures on both sides.
Functional performance | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  Upper limb flexibility will be assessed using the back scratch test. Participants will be instructed to pass one hand over the shoulder and the other from the bottom of the back, trying to reach both hands as close as possible.
Body composition | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  Body composition will be measured through bioelectrical impedance (Impedimed Australia). Data regarding weight, fat mass, lean mass, water percentage, bone mass, visceral fat, and phase angle will be collected from the scale. Participants will be asked to maintain their dietary patterns before the test and refrain from intense exercise the day before. The measurement will be performed under standardized conditions. The height measurement will be considered to the nearest 0.1 cm of the participants and will be performed using a balance-mounted stadiometer (SECA, Germany), with the participants standing and bare-footed. Body weight will be measured to the nearest 0.1kg with a digital scale. BMI (kg/m2) will be calculated from weight (kg) and height (m). Participants will be asked to maintain their dietary patterns before the test and refrain from intense exercise the day before.
Body composition | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  The height measurement will be considered to the nearest 0.1 cm of the participants and will be performed using a balance-mounted stadiometer (SECA, Germany), with the participants standing barefoot.
Body composition | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  Body weight will be measured with a digital scale to the nearest 0.1kg.
Body composition | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  BMI (kg/m2) will be calculated from weight (kg) and height (m).
Physical Activity and Sedentary Behavior | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  PA levels and SB will be assessed using accelerometry (GT9 link, Actigraph). Participants will be instructed to wear the device on an elastic belt on the non-dominant hip for seven days during all waking hours, removing only to sleep. The sampling units (epochs) will be settled to 1s to ease data analysis and ensure the appropriate sensitivity of the device during low-intensity activities. According to specific established thresholds, the accelerometer counts will be categorized into sedentary, light, moderate, and vigorous activity levels. Any interval of 60 or more minutes with continuous zero counts will be considered non-wear time.
Physical Activity and Sedentary Behavior | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  The International Physical Activity Questionnaire Short-Form (IPAQ-SF) comprises nine items that measure the weekly time spent on all intensities PA (i.e., light, moderate, and vigorous) and time spent sitting on week and weekend days. Total PA scores are calculated from the collected data and discriminated by intensity.
General quality of life and breast-cancer specitfic quality of life | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  Quality of life will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30).The EORT QLQ-C30 questionnaire consists of 30 items, grouped into 8 multi-item scales (i.e., functional: physical, role, emotional, cognitive, and social; symptom: fatigue, pain, and nausea), one global health status and quality of life subscale, and 6 single-item questions (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties).
General quality of life and breast-cancer specitfic quality of life | Assessments will be performed at four time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months), 3 month follow-up (throughout the study completion up to 2 years)
  The specific module EORTC QLQ-BR45 will measure breast cancer-related quality of life. The breast cancer module QLQ-BR45 comprises five functional subscales (body image, future perspective, sexual functioning, sexual enjoyment, and breast satisfaction) and seven symptoms subscales (arm symptoms, breast symptoms, endocrine therapy, skin mucositis, endocrine sexual symptoms, systemic therapy side effects, and upset hair loss), for a total of 45 items.

OTHER OUTCOMES:
Demographics | Assessments will be performed at two time points: baseline (throughout recruitment period completion, 1 year), post-intervention (6-12 months)
  Participants' demographic information (e.g., age, education, marital status, and economic status) will be collected through a general information questionnaire
Physical activity history | Assessments will be performed atbaseline (throughout recruitment period completion, 1 year)
  PA history will be collected through a general information questionnaire
Medical history | Assessments will be performed at three time points: baseline (throughout recruitment period completion, 1 year ), mid-treatment (3-6 months), post-intervention (6-12 months)
  Clinical history data will be retrieved from their medical records after they sign the informed consent form.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro B. Júdice, PhD, Study Director — CIDEFES; Eliana V. Carraça, PhD, Study Director — CIDEFES
Locations (1):
- Universidade Lusófona, Centro de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
The corresponding author will make anonymized trial data available for non-commercial research purposes upon reasonable request.
  This trial's findings will be disseminated through publication in leading international oncology scientific journals and presentations at national and international conferences. In addition. the results and mediation analysis will be produced and published. As this is a pragmatic trial with highly applicable outcomes for participants and decision-makers, it presents potential for future widespread implementation through relevant stakeholders.
Supporting Information: Study Protocol
Time Frame: Dissemination policy This trial's findings will be disseminated through publication in leading international oncology scientific journals and presentations at national and international conferences. In addition. the results and mediation analysis will be produced and published. As this is a pragmatic trial with highly applicable outcomes for participants and decision-makers, it presents potential for future widespread implementation through relevant stakeholders.
Access Criteria: The corresponding author will make anonymized trial data available for non-commercial research purposes upon reasonable request.

REFERENCES:
- [Background] Arnold M, Morgan E, Rumgay H, Mafra A, Singh D, Laversanne M, Vignat J, Gralow JR, Cardoso F, Siesling S, Soerjomataram I. Current and future burden of breast cancer: Global statistics for 2020 and 2040. Breast. 2022 Dec;66:15-23. doi: 10.1016/j.breast.2022.08.010. Epub 2022 Sep 2. PMID 36084384
- [Background] Giaquinto AN, Sung H, Miller KD, Kramer JL, Newman LA, Minihan A, Jemal A, Siegel RL. Breast Cancer Statistics, 2022. CA Cancer J Clin. 2022 Nov;72(6):524-541. doi: 10.3322/caac.21754. Epub 2022 Oct 3. PMID 36190501
- [Background] Leidy NK. Functional status and the forward progress of merry-go-rounds: toward a coherent analytical framework. Nurs Res. 1994 Jul-Aug;43(4):196-202. PMID 8047422
- [Background] Tong CKW, Lau B, Davis MK. Exercise Training for Cancer Survivors. Curr Treat Options Oncol. 2020 May 27;21(7):53. doi: 10.1007/s11864-020-00752-w. PMID 32462229
- [Background] Nygren P; SBU-group. Swedish Council on Technology Assessment in Health Care. What is cancer chemotherapy? Acta Oncol. 2001;40(2-3):166-74. doi: 10.1080/02841860151116204. PMID 11441929
- [Background] Kerr AJ, Dodwell D, McGale P, Holt F, Duane F, Mannu G, Darby SC, Taylor CW. Adjuvant and neoadjuvant breast cancer treatments: A systematic review of their effects on mortality. Cancer Treat Rev. 2022 Apr;105:102375. doi: 10.1016/j.ctrv.2022.102375. Epub 2022 Mar 4. PMID 35367784
- [Background] Alfarouk KO, Stock CM, Taylor S, Walsh M, Muddathir AK, Verduzco D, Bashir AH, Mohammed OY, Elhassan GO, Harguindey S, Reshkin SJ, Ibrahim ME, Rauch C. Resistance to cancer chemotherapy: failure in drug response from ADME to P-gp. Cancer Cell Int. 2015 Jul 15;15:71. doi: 10.1186/s12935-015-0221-1. eCollection 2015. PMID 26180516
- [Background] Engle K, Kumar G. Cancer multidrug-resistance reversal by ABCB1 inhibition: A recent update. Eur J Med Chem. 2022 Sep 5;239:114542. doi: 10.1016/j.ejmech.2022.114542. Epub 2022 Jun 17. PMID 35751979
- [Background] Longo DL, Duffey PL, DeVita VT Jr, Wesley MN, Hubbard SM, Young RC. The calculation of actual or received dose intensity: a comparison of published methods. J Clin Oncol. 1991 Nov;9(11):2042-51. doi: 10.1200/JCO.1991.9.11.2042. PMID 1941063
- [Background] Lyman GH, Dale DC, Crawford J. Incidence and predictors of low dose-intensity in adjuvant breast cancer chemotherapy: a nationwide study of community practices. J Clin Oncol. 2003 Dec 15;21(24):4524-31. doi: 10.1200/JCO.2003.05.002. PMID 14673039
- [Background] Wildiers H, Reiser M. Relative dose intensity of chemotherapy and its impact on outcomes in patients with early breast cancer or aggressive lymphoma. Crit Rev Oncol Hematol. 2011 Mar;77(3):221-40. doi: 10.1016/j.critrevonc.2010.02.002. Epub 2010 Mar 15. PMID 20227889
- [Background] Bland KA, Zadravec K, Landry T, Weller S, Meyers L, Campbell KL. Impact of exercise on chemotherapy completion rate: A systematic review of the evidence and recommendations for future exercise oncology research. Crit Rev Oncol Hematol. 2019 Apr;136:79-85. doi: 10.1016/j.critrevonc.2019.02.005. Epub 2019 Feb 16. PMID 30878132
- [Background] Ashcraft KA, Warner AB, Jones LW, Dewhirst MW. Exercise as Adjunct Therapy in Cancer. Semin Radiat Oncol. 2019 Jan;29(1):16-24. doi: 10.1016/j.semradonc.2018.10.001. PMID 30573180
- [Background] Wang Q, Zhou W. Roles and molecular mechanisms of physical exercise in cancer prevention and treatment. J Sport Health Sci. 2021 Mar;10(2):201-210. doi: 10.1016/j.jshs.2020.07.008. Epub 2020 Jul 30. PMID 32738520
- [Background] Zhu C, Ma H, He A, Li Y, He C, Xia Y. Exercise in cancer prevention and anticancer therapy: Efficacy, molecular mechanisms and clinical information. Cancer Lett. 2022 Sep 28;544:215814. doi: 10.1016/j.canlet.2022.215814. Epub 2022 Jul 5. PMID 35803475
- [Background] Kampshoff CS, Jansen F, van Mechelen W, May AM, Brug J, Chinapaw MJ, Buffart LM. Determinants of exercise adherence and maintenance among cancer survivors: a systematic review. Int J Behav Nutr Phys Act. 2014 Jul 2;11:80. doi: 10.1186/1479-5868-11-80. PMID 24989069
- [Background] Sheill G, Guinan E, Brady L, Hevey D, Hussey J. Exercise interventions for patients with advanced cancer: A systematic review of recruitment, attrition, and exercise adherence rates. Palliat Support Care. 2019 Dec;17(6):686-696. doi: 10.1017/S1478951519000312. PMID 31109383
- [Background] Ng AH, Ngo-Huang A, Vidal M, Reyes-Garcia A, Liu DD, Williams JL, Fu JB, Yadav R, Bruera E. Exercise Barriers and Adherence to Recommendations in Patients With Cancer. JCO Oncol Pract. 2021 Jul;17(7):e972-e981. doi: 10.1200/OP.20.00625. Epub 2021 Mar 19. PMID 33739853
- [Background] Mijwel S, Bolam KA, Gerrevall J, Foukakis T, Wengstrom Y, Rundqvist H. Effects of Exercise on Chemotherapy Completion and Hospitalization Rates: The OptiTrain Breast Cancer Trial. Oncologist. 2020 Jan;25(1):23-32. doi: 10.1634/theoncologist.2019-0262. Epub 2019 Aug 7. PMID 31391297
- [Background] Sanft T, Harrigan M, McGowan C, Cartmel B, Zupa M, Li FY, Ferrucci LM, Puklin L, Cao A, Nguyen TH, Neuhouser ML, Hershman DL, Basen-Engquist K, Jones BA, Knobf T, Chagpar AB, Silber A, Tanasijevic A, Ligibel JA, Irwin ML. Randomized Trial of Exercise and Nutrition on Chemotherapy Completion and Pathologic Complete Response in Women With Breast Cancer: The Lifestyle, Exercise, and Nutrition Early After Diagnosis Study. J Clin Oncol. 2023 Dec 1;41(34):5285-5295. doi: 10.1200/JCO.23.00871. Epub 2023 Sep 1. PMID 37656930
- [Background] Denton F, Power S, Waddell A, Birkett S, Duncan M, Harwood A, McGregor G, Rowley N, Broom D. Is It Really Home-Based? A Commentary on the Necessity for Accurate Definitions across Exercise and Physical Activity Programmes. Int J Environ Res Public Health. 2021 Sep 1;18(17):9244. doi: 10.3390/ijerph18179244. PMID 34501833
- [Background] Coughlin SS, Caplan LS, Williams V. Home-based physical activity interventions for breast cancer patients receiving primary therapy: a systematic review. Breast Cancer Res Treat. 2019 Dec;178(3):513-522. doi: 10.1007/s10549-019-05424-4. Epub 2019 Sep 6. PMID 31493034
- [Background] Bates-Fraser LC, Riley S, Stopforth C, Moertl K, Edgar K, Stoner L, Hanson ED. Home-based exercise improves quality of life in breast and prostate cancer survivors: A meta-analysis. PLoS One. 2023 Apr 20;18(4):e0284427. doi: 10.1371/journal.pone.0284427. eCollection 2023. PMID 37079635
- [Background] Ramos PGF, Judice PB, Nobre I, Carraca EV. Home-based exercise interventions' impact on breast cancer survivors' functional performance: a systematic review. J Cancer Surviv. 2025 Aug;19(4):1222-1235. doi: 10.1007/s11764-024-01545-y. Epub 2024 Feb 15. PMID 38356019
- [Background] Dinapoli L, Colloca G, Di Capua B, Valentini V. Psychological Aspects to Consider in Breast Cancer Diagnosis and Treatment. Curr Oncol Rep. 2021 Mar 11;23(3):38. doi: 10.1007/s11912-021-01049-3. PMID 33709235
- [Background] El Kheir DYM, Ibrahim AHM. Epidemiological assessment of distress during chemotherapy: who is affected? J Taibah Univ Med Sci. 2019 Oct 8;14(5):448-453. doi: 10.1016/j.jtumed.2019.08.004. eCollection 2019 Oct. PMID 31728143
- [Background] Ekkekakis P. Let them roam free? Physiological and psychological evidence for the potential of self-selected exercise intensity in public health. Sports Med. 2009;39(10):857-88. doi: 10.2165/11315210-000000000-00000. PMID 19757863
- [Background] Schleicher E, McAuley E, Courneya KS, Anton P, Ehlers DK, Phillips SM, Brown NI, Oster RA, Pekmezi D, Rogers LQ. Breast cancer survivors' exercise preferences change during an exercise intervention are associated with post-intervention physical activity. J Cancer Surviv. 2024 Oct;18(5):1453-1463. doi: 10.1007/s11764-023-01389-y. Epub 2023 Apr 29. PMID 37120460
- [Background] Chen X, Shi X, Yu Z, Ma X. High-intensity interval training in breast cancer patients: A systematic review and meta-analysis. Cancer Med. 2023 Sep;12(17):17692-17705. doi: 10.1002/cam4.6387. Epub 2023 Aug 17. PMID 37587859
- [Background] Ekkekakis P, Biddle SJH. Extraordinary claims in the literature on high-intensity interval training (HIIT): IV. Is HIIT associated with higher long-term exercise adherence? Psychol Sport Exerc. 2023 Jan;64:102295. doi: 10.1016/j.psychsport.2022.102295. Epub 2022 Sep 17. PMID 37665824
- [Background] Ramirez-Parada K, Courneya KS, Muniz S, Sanchez C, Fernandez-Verdejo R. Physical activity levels and preferences of patients with breast cancer receiving chemotherapy in Chile. Support Care Cancer. 2019 Aug;27(8):2941-2947. doi: 10.1007/s00520-018-4595-1. Epub 2018 Dec 18. PMID 30564935
- [Background] Alves RC, Enes A, Follador L, Prestes J, DA Silva SG. Effect of Different Training Programs at Self-Selected Intensity on Body Composition, Perceptual Responses and Fitness Outcomes in Obese Women. Int J Exerc Sci. 2022 Feb 1;15(4):373-385. doi: 10.70252/HJJD8645. eCollection 2022. PMID 36895844
- [Background] Glass SC, Ahmad S, Gabler T. Effectiveness of a 2-Week Strength Training Learning Intervention on Self-selected Weight-Training Intensity. J Strength Cond Res. 2020 Sep;34(9):2443-2448. doi: 10.1519/JSC.0000000000003729. PMID 32732772
- [Background] Ratamess NA, Faigenbaum AD, Hoffman JR, Kang J. Self-selected resistance training intensity in healthy women: the influence of a personal trainer. J Strength Cond Res. 2008 Jan;22(1):103-11. doi: 10.1519/JSC.0b013e31815f29cc. PMID 18296962
- [Background] Power, S., Rowley, N., Duncan, M. & Broom, D. Co-Designing and Refining a Home-Based Exercise Programme for Adults Living with Overweight and Obesity: Insight from People with Lived Experience. Obesities 3, 132-145 (2023).
- [Background] Gildea GC, Spence RR, Jones TL, Turner JC, Macdonald ER, Hayes SC, Sandler CX. Barriers, facilitators, perceptions and preferences influencing physical activity participation, and the similarities and differences between cancer types and treatment stages - A systematic rapid review. Prev Med Rep. 2023 May 24;34:102255. doi: 10.1016/j.pmedr.2023.102255. eCollection 2023 Aug. PMID 37273528
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Kraemer MB, Priolli DG, Reis IGM, Pelosi AC, Garbuio ALP, Messias LHD. Home-based, supervised, and mixed exercise intervention on functional capacity and quality of life of colorectal cancer patients: a meta-analysis. Sci Rep. 2022 Feb 15;12(1):2471. doi: 10.1038/s41598-022-06165-z. PMID 35169171
- [Background] Sharma A, Jasrotia S, Kumar A. Effects of Chemotherapy on the Immune System: Implications for Cancer Treatment and Patient Outcomes. Naunyn Schmiedebergs Arch Pharmacol. 2024 May;397(5):2551-2566. doi: 10.1007/s00210-023-02781-2. Epub 2023 Oct 31. PMID 37906273
- [Background] Courneya KS, Segal RJ, Vallerand JR, Forbes CC, Crawford JJ, Dolan LB, Friedenreich CM, Reid RD, Gelmon K, Mackey JR, McKenzie DC. Motivation for Different Types and Doses of Exercise During Breast Cancer Chemotherapy: a Randomized Controlled Trial. Ann Behav Med. 2016 Aug;50(4):554-63. doi: 10.1007/s12160-016-9782-z. PMID 26896305
- [Background] Winters-Stone KM, Boisvert C, Li F, Lyons KS, Beer TM, Mitri Z, Meyers G, Eckstrom E, Campbell KL. Delivering exercise medicine to cancer survivors: has COVID-19 shifted the landscape for how and who can be reached with supervised group exercise? Support Care Cancer. 2022 Mar;30(3):1903-1906. doi: 10.1007/s00520-021-06669-w. Epub 2021 Nov 6. PMID 34741653
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Borg, G. Borg's Perceived Exertion and Pain Scales. (Human Kinetics, Champaign, IL, 1998).
- [Background] Thorup CB, Gronkjaer M, Spindler H, Andreasen JJ, Hansen J, Dinesen BI, Nielsen G, Sorensen EE. Pedometer use and self-determined motivation for walking in a cardiac telerehabilitation program: a qualitative study. BMC Sports Sci Med Rehabil. 2016 Aug 18;8:24. doi: 10.1186/s13102-016-0048-7. eCollection 2016. PMID 27547404
- [Background] Pudkasam S, Polman R, Pitcher M, Fisher M, Chinlumprasert N, Stojanovska L, Apostolopoulos V. Physical activity and breast cancer survivors: Importance of adherence, motivational interviewing and psychological health. Maturitas. 2018 Oct;116:66-72. doi: 10.1016/j.maturitas.2018.07.010. Epub 2018 Jul 23. PMID 30244781
- [Background] Pudkasam S, Feehan J, Talevski J, Vingrys K, Polman R, Chinlumprasert N, Stojanovska L, Apostolopoulos V. Motivational strategies to improve adherence to physical activity in breast cancer survivors: A systematic review and meta-analysis. Maturitas. 2021 Oct;152:32-47. doi: 10.1016/j.maturitas.2021.06.008. Epub 2021 Jun 24. PMID 34674806
- [Background] Tremblay MS, Aubert S, Barnes JD, Saunders TJ, Carson V, Latimer-Cheung AE, Chastin SFM, Altenburg TM, Chinapaw MJM; SBRN Terminology Consensus Project Participants. Sedentary Behavior Research Network (SBRN) - Terminology Consensus Project process and outcome. Int J Behav Nutr Phys Act. 2017 Jun 10;14(1):75. doi: 10.1186/s12966-017-0525-8. PMID 28599680
- [Background] Cohen, J. Statistical Power Analysis for the Behavioral Sciences. (L. Erlbaum Associates, Hillsdale, N.J, 1988).
- [Background] Kang H. Sample size determination and power analysis using the G*Power software. J Educ Eval Health Prof. 2021;18:17. doi: 10.3352/jeehp.2021.18.17. Epub 2021 Jul 30. PMID 34325496
- [Background] Carraca EV, Rodrigues B, Franco S, Nobre I, Jeronimo F, Ilharco V, Gabriel F, Ribeiro L, Palmeira AL, Silva MN. Promoting physical activity through supervised vs motivational behavior change interventions in breast cancer survivors on aromatase inhibitors (PAC-WOMAN): protocol for a 3-arm pragmatic randomized controlled trial. BMC Cancer. 2023 Jul 5;23(1):632. doi: 10.1186/s12885-023-11137-1. PMID 37407950
- [Background] Hryniuk W, Bush H. The importance of dose intensity in chemotherapy of metastatic breast cancer. J Clin Oncol. 1984 Nov;2(11):1281-8. doi: 10.1200/JCO.1984.2.11.1281. No abstract available. PMID 6387060
- [Background] Van Vulpen JK, Velthuis MJ, Steins Bisschop CN, Travier N, Van Den Buijs BJ, Backx FJ, Los M, Erdkamp FL, Bloemendal HJ, Koopman M, De Roos MA, Verhaar MJ, Ten Bokkel-Huinink D, Van Der Wall E, Peeters PH, May AM. Effects of an Exercise Program in Colon Cancer Patients undergoing Chemotherapy. Med Sci Sports Exerc. 2016 May;48(5):767-75. doi: 10.1249/MSS.0000000000000855. PMID 26694846
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Schmidt K, Vogt L, Thiel C, Jager E, Banzer W. Validity of the six-minute walk test in cancer patients. Int J Sports Med. 2013 Jul;34(7):631-6. doi: 10.1055/s-0032-1323746. Epub 2013 Feb 26. PMID 23444095
- [Background] But-Hadzic J, Dervisevic M, Karpljuk D, Videmsek M, Dervisevic E, Paravlic A, Hadzic V, Tomazin K. Six-Minute Walk Distance in Breast Cancer Survivors-A Systematic Review with Meta-Analysis. Int J Environ Res Public Health. 2021 Mar 5;18(5):2591. doi: 10.3390/ijerph18052591. PMID 33807611
- [Background] Rikli RE, Jones CJ. Development and validation of criterion-referenced clinically relevant fitness standards for maintaining physical independence in later years. Gerontologist. 2013 Apr;53(2):255-67. doi: 10.1093/geront/gns071. Epub 2012 May 20. PMID 22613940
- [Background] Hoenemeyer TW, Cole WW, Oster RA, Pekmezi DW, Pye A, Demark-Wahnefried W. Test/Retest Reliability and Validity of Remote vs. In-Person Anthropometric and Physical Performance Assessments in Cancer Survivors and Supportive Partners. Cancers (Basel). 2022 Feb 21;14(4):1075. doi: 10.3390/cancers14041075. PMID 35205823
- [Background] BECHTOL CO. Grip test; the use of a dynamometer with adjustable handle spacings. J Bone Joint Surg Am. 1954 Jul;36-A(4):820-4; passim. No abstract available. PMID 13174611
- [Background] Huang L, Liu Y, Lin T, Hou L, Song Q, Ge N, Yue J. Reliability and validity of two hand dynamometers when used by community-dwelling adults aged over 50 years. BMC Geriatr. 2022 Jul 15;22(1):580. doi: 10.1186/s12877-022-03270-6. PMID 35840905
- [Background] Polat K, Karadibak D, Guc ZGS, Yavuzsen T, Oztop I. The Relationship between Exercise Capacity and Muscle Strength, Physical Activity, Fatigue and Quality of Life in Patients with Cancer Cachexia. Nutr Cancer. 2024;76(1):55-62. doi: 10.1080/01635581.2023.2276486. Epub 2023 Dec 27. PMID 37917566
- [Background] Rosen B. Recovery of sensory and motor function after nerve repair. A rationale for evaluation. J Hand Ther. 1996 Oct-Dec;9(4):315-27. doi: 10.1016/s0894-1130(96)80037-8. PMID 8994006
- [Background] Paek J, Choi YJ. Association between hand grip strength and impaired health-related quality of life in Korean cancer survivors: a cross-sectional study. BMJ Open. 2019 Sep 8;9(9):e030938. doi: 10.1136/bmjopen-2019-030938. PMID 31501128
- [Background] Esteban-Simon A, Diez-Fernandez DM, Artes-Rodriguez E, Casimiro-Artes MA, Rodriguez-Perez MA, Moreno-Martos H, Casimiro-Andujar AJ, Soriano-Maldonado A. Absolute and Relative Handgrip Strength as Indicators of Self-Reported Physical Function and Quality of Life in Breast Cancer Survivors: The EFICAN Study. Cancers (Basel). 2021 Oct 21;13(21):5292. doi: 10.3390/cancers13215292. PMID 34771456
- [Background] Rikli, R. E. & Jones, C. J. Senior Fitness Test Manual. (Human Kinetics, United Kingdom, 2001).
- [Background] Kolber MJ, Hanney WJ. The reliability and concurrent validity of shoulder mobility measurements using a digital inclinometer and goniometer: a technical report. Int J Sports Phys Ther. 2012 Jun;7(3):306-13. PMID 22666645
- [Background] Yamada Y, Yoshida T, Murakami H, Kawakami R, Gando Y, Ohno H, Tanisawa K, Konishi K, Julien T, Kondo E, Nakagata T, Nanri H, Miyachi M. Phase angle obtained via bioelectrical impedance analysis and objectively measured physical activity or exercise habits. Sci Rep. 2022 Oct 14;12(1):17274. doi: 10.1038/s41598-022-21095-6. PMID 36241873
- [Background] Gil-Herrero L, Pollan M, Martin M, Lopez-Tarruella S, Castellanos M, Casla-Barrio S. The importance of physical exercise in cardiovascular fitness in breast cancer survivors. A cross-sectional study: women in Motion 2.0. Support Care Cancer. 2022 Aug;30(8):6745-6754. doi: 10.1007/s00520-022-06993-9. Epub 2022 May 6. PMID 35524144
- [Background] Khalil SF, Mohktar MS, Ibrahim F. The theory and fundamentals of bioimpedance analysis in clinical status monitoring and diagnosis of diseases. Sensors (Basel). 2014 Jun 19;14(6):10895-928. doi: 10.3390/s140610895. PMID 24949644
- [Background] Cotogni P, Monge T, Fadda M, De Francesco A. Bioelectrical impedance analysis for monitoring cancer patients receiving chemotherapy and home parenteral nutrition. BMC Cancer. 2018 Oct 17;18(1):990. doi: 10.1186/s12885-018-4904-6. PMID 30332998
- [Background] Baharudin, A. et al. Reliability, Technical Error of Measurement and Validity of Height Measurement Using Portable Stadiometer. (2017).
- [Background] Tudor-Locke C, Johnson WD, Katzmarzyk PT. Accelerometer-determined steps per day in US adults. Med Sci Sports Exerc. 2009 Jul;41(7):1384-91. doi: 10.1249/MSS.0b013e318199885c. PMID 19516163
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] Suau Q, Bianchini E, Bellier A, Chardon M, Milane T, Hansen C, Vuillerme N. Current Knowledge about ActiGraph GT9X Link Activity Monitor Accuracy and Validity in Measuring Steps and Energy Expenditure: A Systematic Review. Sensors (Basel). 2024 Jan 26;24(3):825. doi: 10.3390/s24030825. PMID 38339541
- [Background] Bassett DR Jr. Validity and Reliability issues in Objective Monitoring of Physical Activity. Res Q Exerc Sport. 2000 Jun;71 Suppl 2:30-6. doi: 10.1080/02701367.2000.11082783. No abstract available. PMID 25680010
- [Background] Bassett, D. R. & John, D. Use of pedometers and accelerometers in clinical populations: validity and reliability issues. Physical Therapy Reviews 15, 135-142 (2010).
- [Background] Trinh L, Motl RW, Roberts SA, Gibbons T, McAuley E. Estimation of physical activity intensity cut-points using accelerometry in breast cancer survivors and age-matched controls. Eur J Cancer Care (Engl). 2019 Sep;28(5):e13090. doi: 10.1111/ecc.13090. Epub 2019 May 20. PMID 31106924
- [Background] Troiano RP, Berrigan D, Dodd KW, Masse LC, Tilert T, McDowell M. Physical activity in the United States measured by accelerometer. Med Sci Sports Exerc. 2008 Jan;40(1):181-8. doi: 10.1249/mss.0b013e31815a51b3. PMID 18091006
- [Background] Watson KB, Carlson SA, Carroll DD, Fulton JE. Comparison of accelerometer cut points to estimate physical activity in US adults. J Sports Sci. 2014;32(7):660-9. doi: 10.1080/02640414.2013.847278. Epub 2013 Nov 5. PMID 24188163
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Bjelic-Radisic V, Cardoso F, Cameron D, Brain E, Kuljanic K, da Costa RA, Conroy T, Inwald EC, Serpentini S, Pinto M, Weis J, Morag O, Lindviksmoen Astrup G, Tomaszweksi KA, Pogoda K, Sinai P, Sprangers M, Aaronson N, Velikova G, Greimel E, Arraras J, Bottomley A; EORTC Quality of Life Group and Breast Cancer Group. An international update of the EORTC questionnaire for assessing quality of life in breast cancer patients: EORTC QLQ-BR45. Ann Oncol. 2020 Feb;31(2):283-288. doi: 10.1016/j.annonc.2019.10.027. Epub 2019 Dec 18. PMID 31959345
- [Background] Sprangers MA, Groenvold M, Arraras JI, Franklin J, te Velde A, Muller M, Franzini L, Williams A, de Haes HC, Hopwood P, Cull A, Aaronson NK. The European Organization for Research and Treatment of Cancer breast cancer-specific quality-of-life questionnaire module: first results from a three-country field study. J Clin Oncol. 1996 Oct;14(10):2756-68. doi: 10.1200/JCO.1996.14.10.2756. PMID 8874337
- [Background] Tsui TCO, Trudeau M, Mitsakakis N, Torres S, Bremner KE, Kim D, Davis AM, Krahn MD. Developing the Breast Utility Instrument, a preference-based instrument to measure health-related quality of life in women with breast cancer: Confirmatory factor analysis of the EORTC QLQ-C30 and BR45 to establish dimensions. PLoS One. 2022 Feb 4;17(2):e0262635. doi: 10.1371/journal.pone.0262635. eCollection 2022. PMID 35120148
- [Background] Imran M, Al-Wassia R, Alkhayyat SS, Baig M, Al-Saati BA. Assessment of quality of life (QoL) in breast cancer patients by using EORTC QLQ-C30 and BR-23 questionnaires: A tertiary care center survey in the western region of Saudi Arabia. PLoS One. 2019 Jul 10;14(7):e0219093. doi: 10.1371/journal.pone.0219093. eCollection 2019. PMID 31291302
- [Background] Curigliano G, Dunton K, Rosenlund M, Janek M, Cathcart J, Liu Y, Fasching PA, Iwata H. Patient-reported outcomes and hospitalization data in patients with HER2-positive metastatic breast cancer receiving trastuzumab deruxtecan or trastuzumab emtansine in the phase III DESTINY-Breast03 study. Ann Oncol. 2023 Jul;34(7):569-577. doi: 10.1016/j.annonc.2023.04.516. Epub 2023 May 12. PMID 37179020
- [Background] Trewick N, Neumann DL, Hamilton K. Effect of affective feedback and competitiveness on performance and the psychological experience of exercise within a virtual reality environment. PLoS One. 2022 Jun 8;17(6):e0268460. doi: 10.1371/journal.pone.0268460. eCollection 2022. PMID 35675309
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Preacher KJ, Hayes AF. Asymptotic and resampling strategies for assessing and comparing indirect effects in multiple mediator models. Behav Res Methods. 2008 Aug;40(3):879-91. doi: 10.3758/brm.40.3.879. PMID 18697684
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Tunis SR, Stryer DB, Clancy CM. Practical clinical trials: increasing the value of clinical research for decision making in clinical and health policy. JAMA. 2003 Sep 24;290(12):1624-32. doi: 10.1001/jama.290.12.1624. PMID 14506122
- [Background] Lopez P, Galvao DA, Taaffe DR, Newton RU, Souza G, Trajano GS, Pinto RS. Resistance training in breast cancer patients undergoing primary treatment: a systematic review and meta-regression of exercise dosage. Breast Cancer. 2021 Jan;28(1):16-24. doi: 10.1007/s12282-020-01147-3. Epub 2020 Aug 19. PMID 32815096
- [Background] Kjeldsted E, Gehl J, Sorensen DM, Lodin A, Ceballos SG, Dalton SO. Patient-Related Characteristics Associated with Treatment Modifications and Suboptimal Relative Dose Intensity of Neoadjuvant Chemotherapy in Patients with Breast Cancer-A Retrospective Study. Cancers (Basel). 2023 Apr 26;15(9):2483. doi: 10.3390/cancers15092483. PMID 37173949
- [Background] Kanzawa-Lee GA, Larson JL, Resnicow K, Smith EML. Exercise Effects on Chemotherapy-Induced Peripheral Neuropathy: A Comprehensive Integrative Review. Cancer Nurs. 2020 May/Jun;43(3):E172-E185. doi: 10.1097/NCC.0000000000000801. PMID 32187026
- [Background] Schauer T, Hojman P, Gehl J, Christensen JF. Exercise training as prophylactic strategy in the management of neutropenia during chemotherapy. Br J Pharmacol. 2022 Jun;179(12):2925-2937. doi: 10.1111/bph.15141. Epub 2020 Jun 20. PMID 32449810
- [Background] Streckmann F, Balke M, Cavaletti G, Toscanelli A, Bloch W, Decard BF, Lehmann HC, Faude O. Exercise and Neuropathy: Systematic Review with Meta-Analysis. Sports Med. 2022 May;52(5):1043-1065. doi: 10.1007/s40279-021-01596-6. Epub 2021 Dec 29. PMID 34964950
- [Background] Li X, Wang J, Zhang J, Zhang N, Wu C, Geng Z, Zhou J, Dong L. The Effect of Exercise on Weight and Body Composition of Breast Cancer Patients Undergoing Chemotherapy: A Systematic Review. Cancer Nurs. 2023 Jan 16. doi: 10.1097/NCC.0000000000001196. Online ahead of print. PMID 36728172
- [Derived] Ramos PGF, Carraca EV, Valadas G, Batalau RM, Palmeira AL, Silva MN, Viegas PC, Oliveira JG, Pereira SS, Videira-Silva A, Santos IF, Franco S, Gomes D, Teixeira D, Camilo NG, Nobre I, Dias N, Pais J, Koshman D, Judice PB. Home-Combo: an online home-based exercise intervention for women with breast cancer undergoing neoadjuvant chemotherapy: study protocol for a 2-arm pragmatic randomized controlled trial. Front Oncol. 2025 Dec 12;15:1682839. doi: 10.3389/fonc.2025.1682839. eCollection 2025. PMID 41458599

DOCUMENTS (1):
  • Study Protocol (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT06429189/Prot_000.pdf